CLINICAL TRIAL: NCT07005440
Title: Comparison of Functional Training and Dynamic Play Exercise on Gross Motor Skills, Physical Fitness, and Balance in Healthy Children
Brief Title: Functional Training and Dynamic Play Exercise on Gross Motor Skills, Physical Fitness, and Balance in Healthy Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR & AHS/24/0732
Record Dates: First submitted 2025-04-17; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Healthy Children
Keywords: Gross motor skills; Physical fitness; Functional training; Dynamic play exercises; Balance

STUDY DESIGN:
Intervention Model Description: A Randomised clinical trial performed, in which 38 children with the age of 7-10 years will be taken randomly after screening and meeting inclusion criteria.
  Children will be divided in two groups. Group 1 will receive Functional training. This group will receive training a total of 12 week period with one training during 1-8 week and twice a week during 9-12 weeks. Group 2 will receive Dynamic play exercises. This group will receive the lesson once a week during week 1-8 and twice a week during 9-12 weeks. Pre values were taken at baseline and post value will be taken after 12th week of intervention to measure the effects of both therapies.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional Training (Experimental): Group A will perform functional training. Each training session begins with a preparation phase, including warm-up (1-3 min), neuromuscular activation (1-3 min), dynamic stretching (1-3 min), and core muscle activation (1-3 min). The main training phase consists of two modules. The first module is devoted to motor skill development (10-15 mins), with an emphasis on walking, jumping, crawling, throwing, pushing, and catching. The second module focuses on physical fitness (7-10 mins), with an emphasis on balance, agility, and endurance. Each training session concludes with a phase of motor skill consolidation (1-3 min) and static stretching (1-3 min). This group will receive a total 12-week period with one training during 1-8 week and twice a week during 9- 12 weeks
  Interventions: Other: Functional Training; Other: Dynamic Play Exercise
- Dynamic Play Exercise (Active Comparator): Group B will perform dynamic play exercises which includes warm-up (for 3-5 mins), rhythmic exercise (5-10 mins), games (7-10 mins) and free play exercises (10-15 mins). This group will receive the lesson once a week during week 1-8 and twice a week during 9-12 weeks
  Interventions: Other: Functional Training; Other: Dynamic Play Exercise

INTERVENTIONS:
Other: Functional Training — Each training session includes a preparation phase (warm-up, neuromuscular activation, dynamic stretching, and core activation), followed by two main modules: motor skill development (walking, jumping, crawling, throwing, pushing, catching) and physical fitness (balance, agility, endurance). Sessions conclude with motor skill consolidation and static stretching. Training spans 12 weeks: once weekly during weeks 1-8, and twice weekly during weeks 9-12
Other: Dynamic Play Exercise — This includes warm-up (for 3-5 mins), rhythmic exercise (5-10 mins), games (7-10 mins) and free play exercises (10-15 mins). This group will receive the lesson once a week during week 1-8 and twice a week during 9-12 weeks

SUMMARY:
This study aims to explore and compare two distinct approaches to physical activity: functional training and dynamic play exercises, focusing on their effects on children's gross motor skills, physical fitness and balance.

A randomized clinical trial will be conducted. The study will be conducted at Primary school of Lahore in a total duration of 10 months. Sample size will be 38. There will be two groups. Non-probability convenient sampling techniques will be used. The sample having the following characteristics will be included; Age 7-10 years, Both genders, Cognition MMSE score > 25, Class grades 2-5 , BMI between 5th - 85th percentiles, Able to stand and walk independently, PBBS score > 40, TGMD-2 > 13, TUDS > 10 secs. The population having the following characteristics will be excluded from the study; Pes Planus & Pes cavus, Scoliosis, Genu valgum, Genu varum, Juvenile Idiopathic Arthritis, Presence of Asthma, Acute orthopedic problem and any history of surgery past 6 months, visual, vestibular, or balance disorders. The tools that will be included in this study are: Pediatrics balance scale, Test for gross motor development (TGMD-2) and Time up and downstairs test (TUDS). SPSS version 27 will be used for data analyses.

DETAILED DESCRIPTION:
Children's motor development progresses through various milestones such as crawling, walking, and refining fine motor skills, influencing their overall growth and well-being. Piaget's theory underscores the role of motor skills in cognitive and social development, emphasizing that children construct understanding through actions. Motor development, a continuous process, involves gross motor skills (involving large muscles) and fine motor skills (involving small muscles), crucial for daily activities and physical play. Physical fitness in childhood is pivotal for long-term health, correlating with reduced body fat and improved cardio-metabolic health. Balance control, integral to motor skills, depends on sensory inputs and neuromuscular responses. Functional Training and dynamic play are approaches to physical activity that impact gross motor skills, fitness, and balance, with implications for enhancing physical capabilities during childhood. This study aims to explore and compare two distinct approaches to physical activity: functional training and dynamic play exercises, focusing on their effects on children's gross motor skills, physical fitness and balance.

A randomized clinical trial will be conducted. The study will be conducted at Primary school of Lahore in a total duration of 10 months. Sample size will be 38. There will be two groups. Non-probability convenient sampling techniques will be used. The sample having the following characteristics will be included; Age 7-10 years, both genders, cognition MMSE score > 25, Class grades 2-5 , BMI between 5th - 85th percentiles, Able to stand and walk independently, PBBS score > 40, TGMD-2 > 13, TUDS > 10 secs.. The population having the following characteristics will be excluded from the study; Pes Planus & Pes cavus, Scoliosis, Genu valgum, Genu varum, Juvenile Idiopathic Arthritis, Presence of Asthma, Acute orthopedic problem and any history of surgery past 6 months, visual, vestibular, or balance disorders. The tools that will be included in this study are: Pediatrics balance scale, Test for gross motor development (TGMD-2) and Time up and downstairs test (TUDS).

SPSS version 27 will be used for data analyses.

ELIGIBILITY:
Inclusion Criteria:

* Age 7-10 years
* Both genders
* Cognition MMSE score > 25
* Class grades 2-5
* BMI between 5th - 85th percentiles
* Able to stand and walk independently
* PBBS score > 40
* TGMD-2 > 13
* TUDS > 10 secs

Exclusion Criteria:

* Pes Planus & Pes cavus
* Scoliosis
* Genu valgum
* Genu varum
* Juvenile Idiopathic Arthritis
* Presence of Asthma
* Acute orthopedic problem and any history of surgery past 6 months
* Visual, vestibular, or balance disorders

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 38 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2025-07-07 (Estimated); Study Completion 2025-07-07 (Estimated)

PRIMARY OUTCOMES:
Paediatric Balance Scale | Baseline, 12th week
  The Pediatric Balance Scale (PBS), adapted from the Berg Balance Scale, assesses balance in children through 14 items scored 0-4, with a maximum of 56. It shows excellent test-retest (ICC=0.998) and interrater reliability (ICC=0.997).
Test for Gross Motor Development (TGMD-2) | Baseline, 12th week
  The Test of Gross Motor Development-2 (TGMD-2) assesses 12 fundamental movement skills-6 locomotor (e.g., running, hopping) and 6 object control (e.g., throwing, catching)-in children aged 3 to 10 years 11 months. It evaluates movement patterns essential for physical activity. The TGMD-2 shows good internal consistency (α = 0.73-0.87), strong inter-rater agreement (≥ 0.92), and high test-retest reliability (locomotor = 0.91, object control = 0.85).

CONTACTS AND LOCATIONS:
Overall Officials: Zainab Javed, MS-PPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fu T, Zhang D, Wang W, Geng H, Lv Y, Shen R, Bu T. Functional Training Focused on Motor Development Enhances Gross Motor, Physical Fitness, and Sensory Integration in 5-6-Year-Old Healthy Chinese Children. Front Pediatr. 2022 Jul 11;10:936799. doi: 10.3389/fped.2022.936799. eCollection 2022. PMID 35899135